CLINICAL TRIAL: NCT05829915
Title: Feasibility and Efficacy of a Home Exercise Program Using mHealth Technology in People With Parkinson's Disease
Brief Title: mHealth Technology in People With Parkinson's Disease
Acronym: HomTrainPark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Miguel Fernández del Olmo, Proffessor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0801202000720
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Subjects in the intervention group will perform 24 sessions of multisensory training using ROXPro© system (A-Champs)
  Interventions: Device: ROXPro© system (A-Champs)
- Control Group (Active Comparator): Subjects in the Control Group will not perform 24 sessions of multisensory training and they will keep doing the current therapy
  Interventions: Other: No exercise program

INTERVENTIONS:
Device: ROXPro© system (A-Champs) — The intervention consisted in 24 sessions (3/week) of a cognitive-multisensory-physical exercise program carried out in the patient's own home. The exercise program was designed by qualified personal trainers and psychologists, and implemented with the ROXPro© system (A-Champs) (https://a-champs.com; accessed on 8 January 2022). This system consists of small devices that provide visual, auditory and vibration stimuli with which the patient interacts. Through its mobile application, it allows the development of numerous sensory-cognitive-motor exercises adapted to the characteristics of the patients.
  Arms: Intervention Group
Other: No exercise program — The control group did not received the physical exercise program
  Arms: Control Group

SUMMARY:
The main objective of the study is to explore the feasibility and effectiveness of this type of mHalth technology in the treatment of motor symptoms in people with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurological disease whose motor symptoms drastically affect the quality of life of those who suffer from it. There is currently high scientific evidence of the positive effect of physical exercise on the motor function of people with PD. This effect seems to be more relevant when this physical exercise is implemented with external sensory signals (eg visual, auditory). However, the health and socioeconomic context of the patient conditions their access to treatments and physical exercise programs, associationism being common as a low-cost strategy to cover the different therapies. The development of telemedicine, electronic devices and mobile health applications could be an interesting option for those patients who find themselves in the situations mentioned above. However, there are several limitations regarding the use of mobile health apps, such as that less than

1% of them are grounded in research evidence and the digital barrier. Therefore, the main objective of the study is to explore the feasibility and effectiveness of this type of mHalth technology in the treatment of motor symptoms in people with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Absence of treatment with psychotropic drugs or stable dose of the same (without drug or dose modifications in the last four weeks).

In the case of subjects who are part of the intervention group, the following will also be inclusion criteria:

* Caregiver or family member who presents the appropriate skills for collaboration in the implementation of the exercises and in the management of the mobile application.
* Availability of the necessary time for the initial training in the handling of the devices, the development of the sessions and the communication with the researchers.

Exclusion Criteria:

* Insufficient physical condition for participation.
* Sensory deficits that make participation difficult.
* Unstable clinical situation.
* Unstable mental disorder or not adequately controlled with medication (depression, agitation, etc.).
* Presence of associated pathology that involves treatment with drugs that alter cognitive abilities or interfere with the user's participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Speed of gait at preferred pace | baseline
  Speed (m/s)
Speed of gait at preferred pace | at week 8
  Speed (m/s)
Cadence of gait at preferred pace | Baseline
  cadence (steps/min)
Cadence of gait at preferred pace | At week 8
  cadence (steps/min)
Step Length of gait at preferred pace | Baseline
  Step Length (m)
Step Length of gait at preferred pace | At week 8
  Step Length (m)

SECONDARY OUTCOMES:
Time up & go test | Baseline
  Time (seconds)
Time up & go test | At week 8
  Time (seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villamil-Cabello E, Molinero-Martin E, Luque-Casado A, Fernandez-Del-Olmo MA. Home-Based time-constrained reactive training enhances movement speed in upper and lower limbs in Parkinson's disease: A randomized controlled trial. J Parkinsons Dis. 2026 Jan 30:1877718X251405813. doi: 10.1177/1877718X251405813. Online ahead of print. PMID 41615860